CLINICAL TRIAL: NCT03676972
Title: A Prospective, Multi-center, Single-arm Study to Evaluate the Safety and Efficacy of LithoVue Ureteroscope System in Chinese Patients With Urinary Disease(LithoVue China Study)
Brief Title: To Evaluate the Safety and Efficacy of LithoVue Ureteroscope System in Chinese Patients With Urinary Disease
Acronym: LithoVue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U0628
Record Dates: First submitted 2018-07-30; First posted 2018-09-19 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-05

CONDITIONS: Urinary Tract Disease
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LithoVue ureteroscope system (Experimental): The LithoVue System is intended to be used to visualize organs, cavities and canals in the urinary tract (urethra, bladder, ureter, calyces and renal papillae) via transurethral or percutaneous access routes. It can also be used in conjunction with endoscopic accessories to perform various diagnostic and therapeutic procedures in the urinary tract.
  Interventions: Device: LithoVue Ureteroscope System

INTERVENTIONS:
Device: LithoVue Ureteroscope System — The LithoVue System is intended to be used to visualize organs, cavities and canals in the urinary tract (urethra, bladder, ureter, calyces and renal papillae) via transurethral or percutaneous access routes.

SUMMARY:
To evaluate the safety and efficacy of LithoVue ureteroscope system in Chinese population.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, pre-market study.The aim of this study is to evaluate the safety and efficacy of LithoVue ureteroscope system in Chinese population, to support the regulatory approval by CFDA. The study will enroll 60 patients in 3 investigational sites in China. The primary endpoint is procedure success rate of LithoVue ureteroscope system, the procedure success is defined as:Scope condition is suitable to complete the procedure and not requiring immediate scope substitution; it is also considered as a procedure success if the clinical effect is the same as that from the LithoVue scope per investigator's judgement in the case of a scope change (non-LithoVue).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent to participate in the study
2. Willing and able to comply with the study procedures
3. Diagnosed as urinary disease and indicated for flexible ureteroscope procedure
4. For stone cases, the diameter of stones is less than or equal to 2cm in order to avoid staged procedures

Exclusion Criteria:

1. Surgeries are contraindicated
2. Flexible ureterocope procedure is contraindicated
3. Based on doctor's evaluation, the patient's medical condition doesn't fit for this study
4. For stone cases, the diameter of stones is greater than 2cm
5. Women of childbearing potential who are or might be pregnant at the time of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lulin Ma, Doctor, Principal Investigator — Peking University Third Hospital
Locations (3):
- China (3):
  - The First Peking University Hospital, Beijing, Beijing Municipality
  - The Third Peking University Hospital, Beijing, Beijing Municipality
  - Chaoyang Hospital, Beijing, Beijng

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de la Rosette J, Denstedt J, Geavlete P, Keeley F, Matsuda T, Pearle M, Preminger G, Traxer O; CROES URS Study Group. The clinical research office of the endourological society ureteroscopy global study: indications, complications, and outcomes in 11,885 patients. J Endourol. 2014 Feb;28(2):131-9. doi: 10.1089/end.2013.0436. Epub 2013 Dec 17. PMID 24147820
- [Background] Turk C, Petrik A, Sarica K, Seitz C, Skolarikos A, Straub M, Knoll T. EAU Guidelines on Interventional Treatment for Urolithiasis. Eur Urol. 2016 Mar;69(3):475-82. doi: 10.1016/j.eururo.2015.07.041. Epub 2015 Sep 4. PMID 26344917
- [Background] Carey RI, Gomez CS, Maurici G, Lynne CM, Leveillee RJ, Bird VG. Frequency of ureteroscope damage seen at a tertiary care center. J Urol. 2006 Aug;176(2):607-10; discussion 610. doi: 10.1016/j.juro.2006.03.059. PMID 16813899
- [Background] Carey RI, Martin CJ, Knego JR. Prospective evaluation of refurbished flexible ureteroscope durability seen in a large public tertiary care center with multiple surgeons. Urology. 2014 Jul;84(1):42-5. doi: 10.1016/j.urology.2014.01.022. Epub 2014 May 14. PMID 24837456
- [Background] Usawachintachit M, Isaacson DS, Taguchi K, Tzou DT, Hsi RS, Sherer BA, Stoller ML, Chi T. A Prospective Case-Control Study Comparing LithoVue, a Single-Use, Flexible Disposable Ureteroscope, with Flexible, Reusable Fiber-Optic Ureteroscopes. J Endourol. 2017 May;31(5):468-475. doi: 10.1089/end.2017.0027. Epub 2017 Mar 13. PMID 28287823

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LithoVue Ureteroscope System
Started | 60
Completed | 58
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Of the 60 subjects, 54 patients had stones, 5 patients had tumors, and 1 patient had ureteral stricture.
Arm/Group | LithoVue Ureteroscope System
Number analyzed (Participants) | 60
Age, Continuous [Geometric Mean (Standard Deviation); unit: year] | 53.35 (15.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 60
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 60
Body Mass Index (BMI) [Geometric Mean (Standard Deviation); unit: kg/m^2] — Height (cm) and Weight (kg), The formula for BMI is weight in kilograms divided by height in meters squared
  kg/m^2 | 25.21 (4.47)
Indication for flexible ureteroscope procedures [Count of Participants; unit: Participants]
  Tumor | 5
  Stone | 54
  ureteral stricture | 1

OUTCOME MEASURES:

1. Primary Outcome: Procedure Success Rate of LithoVue Ureteroscope System at 4Weeks4Weeks ± 7 Days From Procedure
Description: Procedure success is defined as: Scope condition is suitable to complete the procedure and not requiring immediate scope substitution; it is also considered as a procedure success if the clinical effect is the same as that from the LithoVue scope per investigator's judgement in the case of a scope change (non-LithoVue).
Time Frame: 4Weeks ± 7 days from procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LithoVue Ureteroscope System
Number analyzed (Participants) | 60
percentage of participants | 100 [95.1 to 100]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were assessed the participants in 4 weeks post procedure
Groups:
- All-Cause Mortality and Other AE in Participants Were Assessed for up to 4 Weeks Post Procedure: The LithoVue System is intended to be used to visualize organs, cavities and canals in the urinary tract (urethra, bladder, ureter, calyces and renal papillae) via transurethral or percutaneous access routes. It can also be used in conjunction with endoscopic accessories to perform various diagnostic and therapeutic procedures in the urinary tract.
  LithoVue Ureteroscope System: The LithoVue System is intended to be used to visualize organs, cavities and canals in the urinary tract (urethra, bladder, ureter, calyces and renal papillae) via transurethral or percutaneous access routes.
Arm/Group | All-Cause Mortality and Other AE in Participants Were Assessed for up to 4 Weeks Post Procedure
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-Cause Mortality and Other AE in Participants Were Assessed for up to 4 Weeks Post Procedure (N=60)
Urinary tract infection (Infections and infestations) | 1 (1) — urinary tract infection at four weeks after surgery, which improved after in-patient treatment, then the patient was discharged from the hospital.
Cerebral infarction (Vascular disorders) | 1 (1) — This SAE case was the death of a patient, who died due to acute cerebral infarction 18 days after surgery.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The SAE was sudden dyspnea of a patient during the resuscitation from anesthesia process after the procedure concluded.
Fever (Blood and lymphatic system disorders) | 1 (1) — The SAE was fever, which improved after symptomatic treatment
Fistula rupture (Surgical and medical procedures) | 1 (1) — The SAE was the rupture of the fistula that needed to be indwelled for the discharge of stones after the stone surgery during extubation, and the patient improved after hospitalization during which the remaining fistula in the body was pulled out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT03676972/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03676972/SAP_001.pdf